CLINICAL TRIAL: NCT00785603
Title: Paroxetines Effect on Tramadols Metabolism and Pharmakodynamics: a Dose Response Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Kim Brøsen/ dr. med, Institut of Public Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AKF-374
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Depression; Pain
Keywords: Depression; pain; CYP2D6; interactions; Pupillometry; Tramadol; Paroxetine; MR-ratio
MeSH Terms: conditions — Depression; Pain | interventions — Paroxetine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Paroxetine — tablets of 20 mg paroxetine
  Other Names: Paroxetin, copyfarm
Drug: Paroxetin placebo — capsules with lactulose to hide, whether the volunteer are receiving 0, 10, 20, 30 or 50 mg paroxetine
Drug: Tramadol — Capsules of 50 mg tramadol
  Other Names: Nobligan

SUMMARY:
The purpose of the study is to examine the connection between the dose of paroxetine and the effect of paroxetine on tramadols metabolism and thereby the effect of tramadol on the median pupil size.

In the study 12 healthy volunteers are going through 5 phases where they are suppose to consume a determined dose of tramadol and 5 various doses of paroxetine corresponding to the 5 phases. Fig 1.

phases 1 2 3 4 5 Dosis Tramadol mg 50 50 50 50 50 Dosis Paroxetine mg Placebo 10 20 30 50 Paroxetin / placebo 2 ½ placebo 2 placebo 1 ½ placebo 1 placebo tablets ½ paroxetine 1 paroxetine 1 ½ paroxetine 2 ½ paroxetine Fig. 1 summary of the 5 phases

There is a variation in the time where maximal plasma concentration is obtained in consumption of respectively tramadol (1 - 2 hours) and paroxetine (6 hours). For that reason there has to be at least 6 hours between the administration of paroxetine and tramadol.

The healthy volunteer brings the research medicine home and consumes it before bedtime the night before the day of the study. At eight o'clock next morning the healthy volunteer arrives to the first pupil measurement and consumption of tramadol. Tree hours later the next pupil measurement is carried through. The healthy volunteer accumulates his or her urine until 2 pm. As paroxetine is a irreversible inhibitor of the enzyme CYP2D6 there has to go at least 14 days before the next phase takes place. In that amount of time there can be recreated a new pool of enzyme.

DETAILED DESCRIPTION:
The purpose of the study is to examine the connection between the dose of paroxetine and the effect of paroxetine on tramadols metabolism and thereby the effect of tramadol on the median pupil size.

Tramadol is being metabolized in the liver to O-desmethyltramadol (M1) catalysed by the enzyme P450 CYP2D6 and to N-desmethyltramadol (M2). Tramadol is a racemic mixture of the two enantiomers (+)-tramadol hydrochlorid and (-)-tramadol hydrochlorid and therefore there is formed two enantiomer metabolits, (+)-M1 and (-)-M1. The (+)-M1 has a much higher affinity fore the human opioid µ-receptor compared to (+)-tramadol, (-)-tramadol and (-)-M1.

Paroxetine is a very potent inhibitor of the enzyme CYP2D6 and when there is contemporary administration of paroxetine and tramadol the formation of the active metabolit (+)-M1 will be inhibited. The patient will experience a poorer analgesic effect of tramadol.

It is also the effect of (+)-M1 on the opioid µ-receptor than results in the contracted pupils and that is why it can be shown how potent paroxetine inhibits the enzyme CYP2D6 by measuring the median pupil size.

In the study 12 healthy volunteers are going through 5 phases where they are suppose to consume a determined dose of tramadol and 5 various doses of paroxetine corresponding to the 5 phases. Fig 1.

phases 1 2 3 4 5 Dosis Tramadol mg 50 50 50 50 50 Dosis Paroxetine mg Placebo 10 20 30 50 Paroxetin / placebo 2 ½ placebo 2 placebo 1 ½ placebo 1 placebo tablets ½ paroxetine 1 paroxetine 1 ½ paroxetine 2 ½ paroxetine Fig. 1 summary of the 5 phases

There is a variation in the time where maximal plasma concentration is obtained in consumption of respectively tramadol (1 - 2 hours) and paroxetine (6 hours). For that reason there has to be at least 6 hours between the administration of paroxetine and tramadol.

The healthy volunteer brings the research medicine home and consumes it before bedtime the night before the day of the study. At eight o'clock next morning the healthy volunteer arrives to the first pupil measurement and consumption of tramadol. Tree hours later the next pupil measurement is carried through. The healthy volunteer accumulates his or her urine until 2 pm. As paroxetine is a irreversible inhibitor of the enzyme CYP2D6 there has to go at least 14 days before the next phase takes place. In that amount of time there can be recreated a new pool of enzyme.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers judged from the medical anamnesis and examination, inclusive a laboratory examination.
* Signed written approval and authorization, witch give relevant people (the GCP-unit, the the Danish Medicines Agency and the ethics committee of Southern Denmark) access to documents and data of interest to this study
* Age: 18 - 45 years
* Women must use one of the Danish Medicines Agency defined safe contraception. A negative pregnancy test has to ensure that the volunteers are not pregnant at the start of the study
* All the volunteers have to be phenotyped as CYP2D6 extensive metabolizer (EM) by a "tramadol test": the volunteer ingest 50 mg tramadol and all urine is collected fore 8 hours. By a HPLC method the metabolic ratio (MR) of (-)-M1/(+)-M1 is determined in the urine. Volunteers with a MR-ratio smaller than 2 is defined as CYP2D6 EM's

Exclusion Criteria:

* Any clinical significant observation at the medical- or laboratory examination
* Daily use of medicine or alcohol. Periodic use of medicine can be accepted after individual valuation by a doctor
* Allergy or intolerance to paroxetine or tramadol
* Former participation in a clinical study in the last 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint Pupil measurements Min. diameter mm Reduktion % Latenstime s Maks. constriktions velocity mm/s constriktions velocity mm/s Dilatation velocity mm/s | 3 hours

SECONDARY OUTCOMES:
MR-ratio | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anette Green Nielsen, Stud. pharm, Principal Investigator — Institut of Public Health